CLINICAL TRIAL: NCT04093752
Title: A Randomized, Phase 3, Open-label Trial Comparing the Effect of Tirzepatide Once Weekly Versus Titrated Insulin Glargine on Glycemic Control in Patients With Type 2 Diabetes on Metformin With or Without a Sulfonylurea
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Type 2 Diabetes on Metformin With or Without Sulfonylurea (SURPASS-AP-Combo)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17210; I8F-MC-GPHO (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-09-17; First posted 2019-09-18 (Actual); Results first posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Type 2 Diabetes
Keywords: T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 5 mg Tirzepatide (Experimental): Participants received 5 milligrams (mg) tirzepatide administered subcutaneously (SC) once weekly (QW).
  Interventions: Drug: Tirzepatide
- 10 mg Tirzepatide (Experimental): Participants received 10 mg tirzepatide administered SC QW.
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): Participants received 15 mg tirzepatide administered SC QW.
  Interventions: Drug: Tirzepatide
- Insulin Glargine (Active Comparator): Participants received insulin glargine administered once daily (QD) SC. The starting dose of insulin glargine was 6 Insulin Units (IU)/day at bedtime, titrated to a fasting blood glucose (FBG) between 72-100 milligrams per Deciliter (mg/dL), following a treat-to-target (TTT) algorithm.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 mg Tirzepatide; 15 mg Tirzepatide; 5 mg Tirzepatide
Drug: Insulin Glargine — Administered SC
  Arms: Insulin Glargine

SUMMARY:
The main reason for this study is to compare the study drug tirzepatide to insulin glargine in participants with type 2 diabetes on metformin with or without a sulfonylurea.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Treated with stable metformin with or without a sulfonylurea (metformin ≥1000 milligrams/day; sulfonylurea should be at least half the maximum dose) for at least 2 months
* Are insulin-naive (except for the use of insulin for treatment of gestational diabetes or short-term use [≤14 consecutive days] for acute conditions)
* HbA1c ≥7.5% to ≤11.0% at screening
* Stable weight (±5%) ≥3 months, and agree to not initiate a diet and/or exercise program during the study with the intent of reducing body weight other than the lifestyle and dietary measures for diabetes treatment
* Body mass Index (BMI) ≥23 kilograms per meter squared

Exclusion Criteria:

* Type 1 diabetes mellitus
* Have history of chronic or acute pancreatitis
* Have history of proliferative diabetic retinopathy; or diabetic maculopathy; or non-proliferative diabetic retinopathy that requires acute treatment
* Have a history of severe hypoglycemia and/or hypoglycemia unawareness within the 6 months
* Have a history of ketoacidosis or hyperosmolar state/coma
* Have a known clinically significant gastric emptying abnormality, have undergone or plan to have during the course of the study, or chronically take drugs that directly affect GI motility
* Have acute myocardial infarction (MI), stroke or hospitalization due to congestive heart failure (CHF) within 2 months
* Have family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* Have been treated with prescription drugs that promote weight loss or similar other body weight loss medications including over the counter (OTC) within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 917 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (67):
- Australia (7):
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Illawarra Shoalhaven Local Health District, Wollongong, New South Wales
  - Core Research Group, Milton, Queensland
  - Barwon Health - The Geelong Hospital, Geelong, Victoria
  - Adelaide Medical Solutions, Woodville South
- China (43):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Hebei Medical University, Hengshui Shi, Hebei
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First People's Hospital of Yueyang, Yueyang, Hunan
  - Bao Tou Central Hospital, Baotou, Inner Mongolia
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Hospital of Nanjing, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Medical University - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Dalian University - The Affiliated Zhongshan Hospital, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Shanghai 6th people's hospital, Shanghai, Shanghai Municipality
  - 1st affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Chongqing Three Gorges Central Hospital, Wanzhou, Wanzhou
  - Chongqing General Hospital, Chongqing, Yuzhong District
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Beijing Peking Union Medical College Hospital, Beijing
  - Beijing Pinggu District Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Pingxiang People's Hospital, Pingxiang
  - Shanghai Putuo District Center Hospital, Shanghai
  - Tianjin People's Hospital, Tianjin
  - The Fourth People's Hospital of Zigong City, Zigong
- India (4):
  - King Edward Memorial Hospital and Research Center, Mumbai, Maharashtra
  - BSES Municipal General Hsptl, Mumbai, Maharashtra
  - Apollo Gleneagles Hospitals Kolkata, Kolkata, West Bengal
  - Fortis Hospital, Delhi
- South Korea (13):
  - Kyung Hee University Hospital, Seoul, Gangdong-gu
  - Seoul National University Bundang Hospital, Seongnam, Geonggi-do
  - Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggido
  - Yonsei University Wonju Severance Christian Hospital, Gangwon-do, Korea
  - Ulsan University Hospital, Ulsan, Korea
  - Inje University Sanggye Paik Hospital, Seoul, Seoul-teukbyeolsi
  - Korea University Anam Hospital, Seoul, Seoul-teukbyeolsi
  - Keimyung University Dongsan Hospital, Daegu, Taegu-Kwangyǒkshi
  - Korea University Ansan Hospital, Ansan-si
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Bi Y, Lu S, Tang J, Du L, Ji L. Efficacy and Safety of Tirzepatide in Patients with Type 2 Diabetes: Analysis of SURPASS-AP-Combo by Different Subgroups. Diabetes Ther. 2024 May;15(5):1125-1137. doi: 10.1007/s13300-024-01561-2. Epub 2024 Mar 18. PMID 38494574
- [Derived] Gao L, Lee BW, Chawla M, Kim J, Huo L, Du L, Huang Y, Ji L. Tirzepatide versus insulin glargine as second-line or third-line therapy in type 2 diabetes in the Asia-Pacific region: the SURPASS-AP-Combo trial. Nat Med. 2023 Jun;29(6):1500-1510. doi: 10.1038/s41591-023-02344-1. Epub 2023 May 25. PMID 37231074

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 mg Tirzepatide: Participants received 5 milligrams (mg) tirzepatide administered subcutaneously (SC) once a week (QW).
Period: Overall Study
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Started | 230 | 228 | 229 | 230
Received At Least One Dose of Study Drug | 230 | 228 | 229 | 220
Completed | 213 | 201 | 200 | 201
Not Completed | 17 | 27 | 29 | 29
Not completed — Adverse Event | 7 | 19 | 18 | 4
Not completed — Withdrawal by Subject | 6 | 6 | 8 | 20
Not completed — Lost to Follow-up | 2 | 1 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 2
Not completed — Participant Could Not Continue Due to Work Related Reasons | 0 | 1 | 0 | 1
Not completed — Covid 19 | 0 | 0 | 0 | 1
Not completed — Participant Thought there were Too Many Adverse Events | 0 | 0 | 1 | 0
Not completed — Participant was Reluctant to Follow-up | 1 | 0 | 0 | 0
Not completed — Participant Did Not Come for the Visit | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- 5 mg Tirzepatide: Participants received 5 mg tirzepatide administered SC QW.
- Insulin Glargine: Participants received insulin glargine administered QD SC. The starting dose of insulin glargine was 6 IU/day at bedtime, titrated to a FBG between 72-100 mg/dL, following a TTT algorithm.
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine | Total
Number analyzed (Participants) | 230 | 228 | 229 | 220 | 907
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.10 (11.25) | 53.50 (11.14) | 54.30 (11.65) | 55.60 (11.40) | 54.10 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 102 | 100 | 102 | 400
  Male | 134 | 126 | 129 | 118 | 507
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 230 | 228 | 229 | 220 | 907
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 225 | 225 | 226 | 216 | 892
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 3 | 0 | 5
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 0 | 4 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 5 | 3 | 3 | 4 | 15
  China | 190 | 192 | 190 | 184 | 756
  India | 9 | 7 | 9 | 7 | 32
  South Korea | 26 | 26 | 27 | 25 | 104
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.77 (0.976) | 8.70 (0.955) | 8.67 (0.960) | 8.68 (0.934) | 8.71 (0.956)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Hemoglobin A1c (HbA1c) (10 mg and 15 mg)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed model repeated measures (MMRM) model with covariates Baseline + Country + Baseline Oral Antihyperglycemic Medication (OAM) Use (Metformin (Met), Met plus Sulfonylurea (SU)) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: All randomized participants belonging to the 10 mg, 15 mg Tirzepatide and Insulin Glargine arms who received at least one dose of study drug, had a baseline and at least one post-baseline value, excluding data after initiating rescue antihyperglycemic medication or stopping study drug (last dose date + 7 days).
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 194 | 193 | 193
Percentage of HbA1c | -2.44 (0.073) | -2.49 (0.072) | -0.95 (0.073)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Test type: Non-Inferiority — The study was powered for superiority in HbA1c. The sample size provided >99% power to show noninferiority assuming a 0.4% noninferiority (NI) boundary, 0.45% greater mean reduction in tirzepatide doses compared to insulin glargine, 1:1:1:1 randomization, a common standard deviation (SD) of 1.2%, one-sided significance level of 0.0125 and a dropout rate of 25%; LS Mean Difference = -1.49, 95% CI 2-sided [-1.69 to -1.29]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Test type: Non-Inferiority — The study was powered for superiority in HbA1c. The sample size provided >99% power to show noninferiority assuming a 0.4% NI boundary, 0.45% greater mean reduction in tirzepatide doses compared to insulin glargine, 1:1:1:1 randomization, a common SD of 1.2%, one-sided significance level of 0.0125 and a dropout rate of 25%; LS Mean Difference = -1.54, 95% CI 2-sided [-1.74 to -1.34]

2. Secondary Outcome: Mean Change From Baseline in HbA1c (5 mg)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. LS mean was determined by MMRM model with covariates Baseline + Country + Baseline OAM Use (Met, Met plus SU) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: All randomized participants belonging to the 5 mg Tirzepatide and Insulin Glargine arms who received at least one dose of study drug, had a baseline and at least one post-baseline value, excluding data after initiating rescue antihyperglycemic medication or stopping study drug (last dose date + 7 days).
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 5 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 211 | 193
Percentage of HbA1c | -2.24 (0.070) | -0.95 (0.073)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; LS Mean Difference = -1.29, 95% CI 2-sided [-1.49 to -1.09]

3. Secondary Outcome: Mean Change From Baseline in Body Weight
Description: LS mean was determined by MMRM model with Baseline + Country + Baseline OAM Use (Met, Met plus SU) + Baseline HbA1c Group (<= 8.5%, >8.5%) + Treatment + Time + Treatment*Time (Type III sum of squares) as covariates.
Time Frame: Baseline, Week 40
Population: All randomized participants who received at least one dose of study drug, had a baseline and at least one post-baseline value, excluding data after initiating rescue antihyperglycemic medication or stopping study drug (last dose date + 7 days).
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 211 | 194 | 193 | 194
kilograms (kg) | -5.0 (0.32) | -7.0 (0.33) | -7.2 (0.33) | 1.5 (0.33)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -6.5, 95% CI 2-sided [-7.4 to -5.6]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -8.5, 95% CI 2-sided [-9.5 to -7.6]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -8.7, 95% CI 2-sided [-9.6 to -7.7]

4. Secondary Outcome: Percentage of Participants Achieving an HbA1c Target Value of <7.0%
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Imputed data includes observed value and imputed value if endpoint measure is missing.
Time Frame: Week 40
Population: All randomized participants who received at least one dose of study drug and had a baseline and at least one post-baseline value, excluding data after initiating rescue antihyperglycemic medication or stopping study drug (last dose date + 7 days).
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 228 | 222 | 224 | 215
Percentage of participants | 75.44 | 86.04 | 84.38 | 23.72
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 14.54, 95% CI 2-sided [8.94 to 23.64]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 28.76, 95% CI 2-sided [16.72 to 49.49]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 25.27, 95% CI 2-sided [14.88 to 42.95]

5. Secondary Outcome: Percentage of Participants Achieving an HbA1c Target Value of <5.7%
Description: HbA1c is the glycosylated fraction of hemoglobin A. Imputed data includes observed value and imputed value if endpoint measure is missing.
Time Frame: Week 40
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 228 | 222 | 224 | 215
Percentage of participants | 14.91 | 20.72 | 27.68 | 0.00
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 82.54, 95% CI 2-sided [5.13 to 1327.81]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 124.76, 95% CI 2-sided [7.79 to 1997.01]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 184.90, 95% CI 2-sided [11.59 to 2950.73]

6. Secondary Outcome: Mean Change From Baseline in Fasting Serum Glucose
Description: Fasting serum glucose (FSG) is a test to determine sugar levels in serum sample after an overnight fast. LS mean was determined by MMRM model with Baseline + Country + Baseline OAM Use (Met, Met plus SU) + Baseline HbA1c Group (<= 8.5%, >8.5%) + Treatment + Time + Treatment*Time (Type III sum of squares) as covariates.
Time Frame: Baseline, Week 40
Population: All randomized participants who had received at least one dose of study drug, had a baseline and at least one post-baseline value, excluding data after initiating rescue antihyperglycemic medication or stopping study drug (last dose date + 7 days).
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 206 | 193 | 192 | 194
milligrams per deciliter (mg/dL) | -58.6 (2.13) | -66.2 (2.19) | -64.8 (2.19) | -46.2 (2.19)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -12.3, 95% CI 2-sided [-18.3 to -6.3]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -20.0, 95% CI 2-sided [-26.1 to -13.9]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -18.6, 95% CI 2-sided [-24.6 to -12.5]

7. Secondary Outcome: Mean Change in Daily Glucose Average From Baseline in 7-Point Self-Monitored Blood Glucose (SMBG) Values
Description: The SMBG data was collected at the following 7 time points: Morning Premeal - Fasting, Morning 2-hour Post-meal, Midday Premeal, Midday 2-hour Post-meal, Evening Premeal, Evening 2-hour Post-meal and Bedtime. LS mean was determined by MMRM model with Baseline + Country + Baseline OAM Use (Met, Met plus SU) + Baseline HbA1c Group (<= 8.5%, >8.5%) + Treatment + Time + Treatment*Time (Type III sum of squares) as covariates.
Time Frame: Baseline, Week 40
Population: All randomized participants who have received at least one dose of study drug, had a baseline and at least one post-baseline value, excluding data after initiating rescue antihyperglycemic medication or stopping study drug (last dose date + 7 days).
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 204 | 193 | 186 | 188
milligrams per deciliter (mg/dL) | -77.0 (2.09) | -83.4 (2.16) | -84.6 (2.18) | -42.8 (2.18)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -34.2, 95% CI 2-sided [-40.1 to -28.3]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -40.6, 95% CI 2-sided [-46.7 to -34.6]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -41.8, 95% CI 2-sided [-47.9 to -35.8]

8. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss ≥5%
Description: Imputed data includes observed value and imputed value if endpoint measure is missing.
Time Frame: Week 40
Population: All randomized participants who received at least one dose of study drug, had a baseline and had at least one post-baseline value, excluding data after initiating rescue antihyperglycemic medication or stopping study drug (last dose date + 7 days).
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 228 | 222 | 224 | 215
Percentage of participants | 55.70 | 71.62 | 74.11 | 5.58
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 21.89, 95% CI 2-sided [11.63 to 41.20]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 43.79, 95% CI 2-sided [22.96 to 83.50]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 48.41, 95% CI 2-sided [25.34 to 92.49]

9. Secondary Outcome: Diabetes Treatment Satisfaction as Measured by the Diabetes Treatment Satisfaction Questionnaire, Change Version (DTSQc) Hyperglycemia, Hypoglycemia and Treatment Satisfaction Score
Description: DTSQc, an 8-item questionnaire, assesses relative change in treatment satisfaction perceived frequency of hyperglycemia, and perceived frequency of hypoglycemia from baseline to week 40 or early termination. The treatment satisfaction score ranges from -18 to 18 where the higher the score the greater the improvement in satisfaction with treatment. The lower the score the greater the deterioration in satisfaction with treatment. The hyperglycemia and hypoglycemia scores range from -3 to 3 where negative scores indicate fewer problems with blood glucose levels and positive scores indicate more problems than before. LS mean was determined by ANCOVA model for endpoint measures with Baseline + Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Baseline OAM Use (Met, Met plus SU) + Treatment (Type III sum of squares) as covariates.
Time Frame: Baseline, Week 40
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 212 | 200 | 195 | 196
Units on a scale
  Hyperglycemia | -1.8 (0.12) | -2.1 (0.12) | -2.0 (0.12) | -1.3 (0.12)
  Hypoglycemia | -1.9 (0.11) | -1.9 (0.12) | -2.0 (0.12) | -1.8 (0.12)
  Treatment Satisfaction Score | 16.0 (0.27) | 15.8 (0.28) | 15.9 (0.29) | 14.2 (0.28)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Hyperglycemia; Test type: Superiority; p = 0.007, ANCOVA; LS Mean Difference = -0.47, 95% CI 2-sided [-0.81 to -0.13]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Hyperglycemia; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.77, 95% CI 2-sided [-1.11 to -0.43]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Hyperglycemia; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.71, 95% CI 2-sided [-1.05 to -0.36]
Statistical Analysis 4: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Hypoglycemia; Test type: Superiority; p = 0.384, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.46 to 0.18]
Statistical Analysis 5: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Hypoglycemia; Test type: Superiority; p = 0.307, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.49 to 0.16]
Statistical Analysis 6: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Hypoglycemia; Test type: Superiority; p = 0.184, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.55 to 0.11]
Statistical Analysis 7: Comparison: 5 mg Tirzepatide vs Insulin Glargine; Treatment Satisfaction Score; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 1.81, 95% CI 2-sided [1.03 to 2.59]
Statistical Analysis 8: Comparison: 10 mg Tirzepatide vs Insulin Glargine; Treatment Satisfaction Score; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 1.63, 95% CI 2-sided [0.84 to 2.41]
Statistical Analysis 9: Comparison: 15 mg Tirzepatide vs Insulin Glargine; Treatment Satisfaction Score; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 1.68, 95% CI 2-sided [0.89 to 2.47]

10. Secondary Outcome: Rate of Hypoglycemia With Blood Glucose < 54 mg/dL or Severe Hypoglycemia
Description: The hypoglycemia events were defined by participant reported events with blood glucose < 54 mg/dL [<3.0 Millimole per Liter (mmol/L)] or severe hypoglycemia. Severe hypoglycemia is defined as an episode with severe cognitive impairment requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. The rate of post-baseline hypoglycemia was estimated by negative binomial model: Number of episodes = Country + Baseline OAM Use (Met, Met plus SU) + Baseline HbA1c Group (<= 8.5%, >8.5%) + Treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Baseline through end of safety follow-up (Up To Week 44)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Episodes/participant/365.25 days
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
Number analyzed (Participants) | 230 | 228 | 229 | 220
Episodes/participant/365.25 days | 0.0658 (0.02603) | 0.0890 (0.03196) | 0.0700 (0.02273) | 0.0538 (0.01594)

ADVERSE EVENTS:
Time Frame: Baseline Through End of Safety Follow-Up (Up To Week 44).
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Glargine
All-Cause Mortality (participants affected / at risk) | 0/230 | 0/228 | 1/229 | 2/220
Serious Adverse Events (participants affected / at risk) | 15/230 | 14/228 | 15/229 | 20/220
Other Adverse Events (participants affected / at risk) | 174/230 | 201/228 | 193/229 | 83/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=230) | 10 mg Tirzepatide (N=228) | 15 mg Tirzepatide (N=229) | Insulin Glargine (N=220)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0/134 (0) | 0/126 (0) | 0/129 (0) | 1/118 (1)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac function test (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian germ cell teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/96 (0) | 0/102 (0) | 1/100 (1) | 0/102 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/96 (1) | 0/102 (0) | 0/100 (0) | 0/102 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0/96 (0) | 0/102 (0) | 0/100 (0) | 1/102 (1)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide (N=230) | 10 mg Tirzepatide (N=228) | 15 mg Tirzepatide (N=229) | Insulin Glargine (N=220)
Abdominal distension (Gastrointestinal disorders) | 19 (54) | 25 (63) | 34 (73) | 2 (2)
Constipation (Gastrointestinal disorders) | 12 (13) | 17 (23) | 23 (33) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 77 (181) | 103 (277) | 101 (301) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 6 (32) | 11 (15) | 12 (38) | 3 (4)
Eructation (Gastrointestinal disorders) | 10 (19) | 14 (47) | 9 (35) | 0 (0)
Flatulence (Gastrointestinal disorders) | 20 (40) | 23 (70) | 18 (52) | 2 (2)
Nausea (Gastrointestinal disorders) | 46 (100) | 75 (230) | 73 (231) | 5 (6)
Vomiting (Gastrointestinal disorders) | 21 (32) | 34 (105) | 29 (79) | 3 (4)
Asthenia (General disorders) | 7 (8) | 14 (17) | 10 (13) | 1 (1)
Fatigue (General disorders) | 12 (14) | 23 (44) | 17 (36) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 16 (17) | 14 (18) | 14 (19) | 17 (21)
Amylase increased (Investigations) | 12 (15) | 16 (19) | 15 (17) | 4 (4)
Lipase increased (Investigations) | 32 (36) | 32 (34) | 30 (35) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 74 (179) | 109 (331) | 102 (259) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (12) | 2 (2) | 2 (4) | 18 (27)
Hyperlipidaemia (Metabolism and nutrition disorders) | 7 (7) | 8 (8) | 9 (9) | 11 (11)
Hyperuricaemia (Metabolism and nutrition disorders) | 27 (28) | 28 (35) | 27 (28) | 24 (27)
Dizziness (Nervous system disorders) | 10 (16) | 13 (21) | 24 (37) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT04093752/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT04093752/SAP_001.pdf